CLINICAL TRIAL: NCT01618942
Title: To Measure Pain Perception With Electronic Pressure Algometer of Different Size Probes : a Healthy Subjects Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xianwei Zhang (Other)
Responsible Party: Sponsor-Investigator, Xianwei Zhang, Clinical Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: Pressure algometer
Record Dates: First submitted 2012-06-12; First posted 2012-06-13 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- male subjects (Experimental): grouped by gender and applied pressure pain test
  Interventions: Device: pressure algometer
- female subjects (Experimental): grouped by gender and applied pressure pain test
  Interventions: Device: pressure algometer

INTERVENTIONS:
Device: pressure algometer

SUMMARY:
This study was conducted to explore the influencing factors, subjects and testers' evaluation about pain measurement with hand-held pressure algometer with different size probes. Methods:100 healthy undergraduate students(50 males and 50 females) were recruited into this study. Pain measurement including pressure pain threshold (PPT) and pressure pain tolerance(PTO) was carried out by the hand-held pressure algometer with different size probes (from 1cm2 to 0.01cm2) on three different measuring spots in right forearm. We recorded subjects' skinfold thickness, time per test procedure, types of pain perception, receptivity and degree of accuracy as well as testers' level of laborious.

DETAILED DESCRIPTION:
Subjects with the following diseases were excluded: known history of chronic disease, psychiatric diseases or communication disorders, diabetes mellitus, severe cardiovascular diseases, kidney or liver diseases with poor hepatic function, alcohol or drug abuse, heavy smoker, Pregnancy or at lactation period .

ELIGIBILITY:
Inclusion Criteria:

Aged 20 to 30 The right hand is handedness Agreed to participate the research Not with known chronic disease Not taking analgesics within 3 months

Exclusion Criteria:

* History of chronic pain Psychiatric diseases Diabetes mellitus Severe cardiovascular diseases Kidney or liver diseases Alcohol or drug abuse Heavy smoker Disagree to participate to the research

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Xianwei, Doctor, Study Director — Huazhong University of Science and Technology
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From June 2012 to December 2012, 100 health students were recruitmented in the Tongji Medical College, Huazhong University of Science&Technology, Wuhan China.
Pre-assignment Details: There was no significant events and approaches for the overall study.
Groups:
- Male Subjects: grouped by gender and applied with hand-held pressure algometer with differen
- Female Subjects: grouped by gender grouped by gender and applied with hand-held pressure algometer with differen
Period: Overall Study
Arm/Group | Male Subjects | Female Subjects
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Male Subjects; Female Subjects: grouped by gender
- Total: Total of all reporting groups
Arm/Group | Male Subjects | Female Subjects | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (1.3) | 24.2 (1.9) | 24.2 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 50 | 50
  Male | 50 | 0 | 50
Region of Enrollment [Number; unit: participants]
  China | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Pressure Pain Threshold (PPT)With 1 cm2 Probe
Description: The value was calculated as a avarage value of different measurement sites
Time Frame: 1 hour after the procedure
Measure: Mean (Standard Deviation); unit: kg/cm2
Arm/Group | Male Subjects | Female Subjects
Number analyzed (Participants) | 50 | 50
kg/cm2 | 2.61 (0.88) | 2.20 (0.73)

2. Secondary Outcome: Time of Each Test Procedure
Time Frame: 10 minutes after the procedure
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Male Subjects | Female Subjects
Number analyzed (Participants) | 50 | 50
seconds | 16.8 (5.3) | 14.2 (4.9)

3. Secondary Outcome: Measuring Values of Skinfold Thickness
Time Frame: 10 minutes after the procedure
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Male Subjects | Female Subjects
Number analyzed (Participants) | 50 | 50
millimeters | 3.4 (1.1) | 4.3 (1.3)

4. Primary Outcome: Pressure Pain Tolerance (PTO) With 1cm2 Probe
Description: The value was calculated as a avarage value of different measurement sites
Time Frame: 1 hour after the procedure
Measure: Mean (Standard Deviation); unit: kg/cm2
Arm/Group | Male Subjects | Female Subjects
Number analyzed (Participants) | 50 | 50
kg/cm2 | 5.13 (1.79) | 4.39 (1.52)

5. Primary Outcome: Pressure Pain Threshold (PPT)With 0.1 cm2 Probe
Description: The value was calculated as a avarage value of different measurement sites
Time Frame: 1 hour after the procedure
Measure: Mean (Standard Deviation); unit: kg/cm2
Arm/Group | Male Subjects | Female Subjects
Number analyzed (Participants) | 50 | 50
kg/cm2 | 1.61 (0.71) | 1.11 (0.49)

6. Primary Outcome: Pressure Pain Threshold (PPT)With 0.01 cm2 Probe
Description: The value was calculated as a avarage value of different measurement sites
Time Frame: 1 hour after the procedure
Measure: Mean (Standard Deviation); unit: kg/cm2
Arm/Group | Male Subjects | Female Subjects
Number analyzed (Participants) | 50 | 50
kg/cm2 | 0.45 (0.16) | 0.44 (0.23)

7. Primary Outcome: Pressure Pain Tolerance (PTO) With 0.1cm2 Probe
Description: The value was calculated as a avarage value of different measurement sites
Time Frame: 1 hour after the procedure
Measure: Mean (Standard Deviation); unit: kg/cm2
Arm/Group | Male Subjects | Female Subjects
Number analyzed (Participants) | 50 | 50
kg/cm2 | 3.19 (1.16) | 2.34 (0.90)

8. Primary Outcome: Pressure Pain Tolerance (PTO) With 0.01cm2 Probe
Description: The value was calculated as a avarage value of different measurement sites
Time Frame: 1 hour after the procedure
Measure: Mean (Standard Deviation); unit: kg/cm2
Arm/Group | Male Subjects | Female Subjects
Number analyzed (Participants) | 50 | 50
kg/cm2 | 0.92 (0.32) | 0.93 (0.39)

ADVERSE EVENTS:
Arm/Group | Male Subjects | Female Subjects
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
There was no significant limitation in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No